CLINICAL TRIAL: NCT04067674
Title: Evaluation of Immunosuppression in Septic Shock: Biomarkers and Pharmacological Restoration
Brief Title: Septic Shock-induced Immunosuppression
Acronym: IMMUNOSEPSIS 4
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0071
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic shock patients: Patients included in this cohort will have blood sampling for measurement of immune related biomarkers (immunophenotyping, functional tests, messenger ribonucleic acid (mRNA), circulating markers) in circulating blood and their associations with relevant clinical outcomes
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood sampling for biomarker measurement

SUMMARY:
Septic syndromes are a major although largely under-recognized health care problem and represent the first cause of mortality in intensive care units (ICU). While it has long been known that sepsis deeply perturbs immune homeostasis by inducing a tremendous systemic inflammatory response, novel findings indicate that sepsis indeed initiates a more complex immune response that varies over time, with the concomitant occurrence of both pro- and anti-inflammatory mechanisms. As a resultant, after a short pro-inflammatory phase, septic patients enter a stage of protracted immunosuppression. This is illustrated in those patients by reactivation of dormant viruses (cytomegalovirus (CMV) or Herpes Simplex Virus (HSV)) or infections due to pathogens, including fungi, which are normally pathogenic solely in immunocompromised hosts. These alterations might be directly responsible for worsening outcome in patients who survived initial resuscitation as nearly all immune functions are deeply compromised. New promising therapeutic strategies are currently emerging from those recent findings such as adjunctive immunostimulation for the most immunosuppressed patients. The prerequisite for immunostimulation administration (Interferon gama (IFNg), Granulocyte Macrophage Colony Stimulating Factor (GM-CSF), interleukin 7 (IL-7)) however relies on clinicians' capacity to identify patients who could benefit the most from these immunoadjuvant therapies, as there is no clinical sign of immune dysfunctions.

In this context, the main objectives of IMMUNOSEPSIS 4 study are:

1. to identify the best biomarkers for sepsis-induced immunosuppression
2. to evaluate ex vivo candidate treatments which could rejuvenate immune functions after septic shock

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patient admitted to ICU
* Diagnosis of septic shock within less than 48h at time of screening defined by :
* Presence of a microbiologically diagnosed or suspected infection
* Initiation of a vasopressive treatment to maintain mean arterial blood pressure ≥ 65 mm Hg initiated during the first 48h after ICU admission
* Presence of an hyperlactatemia > 2 mmol/L (18 mg/dL) during the 24h before or after initiation of vasopressive treatment despite adequate volemic reanimation (30 ml/kg)
* Blood sample at D3/D4 available (lab working days)
* Non opposition to study participation obtained from patient or next of kin

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient with no social security insurance, with restricted liberty or under legal protection
* Language barrier
* Patient taking part in interventional study about medicin that could interfere with biologic results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock
Sampling Method: Non-Probability Sample
Enrollment: 305 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2024-11-21 (Estimated); Study Completion 2024-11-21 (Estimated)

PRIMARY OUTCOMES:
Major Histocompatibility Complex (MHC) class II expression rate | at day 3 post septic shock diagnosis
  Association between decreased MHC class II expression on monocytes at day 3 post diagnosis and occurrence of secondary ICU-acquired infections

SECONDARY OUTCOMES:
ICU-acquired infections occurence | 28 days post septic shock diagnosis
  Association between decreased MHC class II expression on monocytes at day 3 post diagnosis and occurrence of secondary Intensive Care Unit (ICU)-acquired infections
mortality rate | 28 days post septic shock diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne VENET, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Venet M, Bidar F, Derive M, Delwarde B, Monard C, Hengy B, Jolly L, Rimmele T, Lukaszewicz AC, Monneret G, Venet F. Persistently Elevated Soluble Triggering Receptor Expressed on Myeloid Cells 1 and Decreased Monocyte Human Leucocyte Antigen DR Expression Are Associated With Nosocomial Infections in Septic Shock Patients. Crit Care Explor. 2023 Feb 24;5(3):e0869. doi: 10.1097/CCE.0000000000000869. eCollection 2023 Mar. PMID 36861044
- [Derived] Coudereau R, Gossez M, Py BF, Henry T, Lukaszewicz AC, Monneret G, Venet F. Monitoring NLRP3 Inflammasome Activation and Exhaustion in Clinical Samples: A Refined Flow Cytometry Protocol for ASC Speck Formation Measurement Directly in Whole Blood after Ex Vivo Stimulation. Cells. 2022 Oct 20;11(20):3306. doi: 10.3390/cells11203306. PMID 36291172